CLINICAL TRIAL: NCT04748029
Title: Evaluation of the Prognostic Role of the Systemic Immune Inflammation Index in Postmenopausal Osteoporosis
Status: Completed | Type: Observational
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Elzem Bolkan Günaydın, Lecturer Doctor, Ufuk University
Other Study IDs: 2020-4-26
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Osteoporosis, Postmenopausal; Osteoporotic Fractures
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporotic Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Systemic immune inflammation index — The systemic immune inflammation index (SII) was calculated using the formula, SII = platelet count x neutrophil count / lymphocyte count. Systemic immune inflammation index (SII) is a new index related to systemic inflammation calculated by the numbers of lymphocytes, neutrophils and platelets in peripheral blood.

SUMMARY:
This study is a retrospective case-control study. In the study, the data of 304 patients who were evaluated in our clinic between January 2017 and January 2020 with a pre-diagnosis or diagnosis of postmenopausal osteoporosis were retrospectively reviewed. Lumbar 1-4 and femoral neck bone mineral densitometry values T scores, ages, sedimentation, C-reactive protein, neutrophil, leukocyte and platelet levels, and mean platelet volume values of the patients were recorded. The neutrophil-lymphocyte ratio was calculated by dividing the neutrophil count by the lymphocyte count, and the platelet-lymphocyte ratio was calculated by dividing the platelet count by the lymphocyte count. The systemic immune inflammation index (SII) was calculated using the formula, SII = platelet count x neutrophil count / lymphocyte count. The aim of this study is to evaluate the prognostic value of the systemic immune inflammation index in postmenopausal osteoporosis and to examine the SII, N / L, PLT / L, MPV, sedimentation (ESR), C reactive protein (CRP), femur and lumbar BMD values and their relationships with each other.

ELIGIBILITY:
Inclusion Criteria:

* Having applied to our clinic with the diagnosis or pre-diagnosis of postmenopausal osteoporosis or osteoporosis with pathological fractures

Exclusion Criteria:

* Having a diagnosis of osteoporosis due to conditions other than postmenopausal osteoporosis
* Those with acute or chronic infection, malignancy and systemic diseases that may change the hematological inflammation parameters to be checked
* Persons who are missing one or more of the parameters planned to be considered among the obtained data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the study, the data of 139 patients who were evaluated in our clinic between January 2017 and January 2020 with a pre-diagnosis or diagnosis of postmenopausal osteoporosis were retrospectively reviewed.
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Systemic immune inflammation index (SII) | 1 month
  Systemic immune inflammation index (SII) is a new index related to systemic inflammation calculated by the numbers of lymphocytes, neutrophils and platelets in peripheral blood defined in 2014. The systemic immune inflammation index (SII) is calculated using the formula, SII = platelet count x neutrophil count / lymphocyte count.

CONTACTS AND LOCATIONS:
Locations (1):
- Ufuk University, Ankara, Çankaya, Turkey (Türkiye)